CLINICAL TRIAL: NCT03223493
Title: Awareness, Care & Treatment in Obesity Management (ACTION) Study
Acronym: ACTION
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-4409; U1111-1198-9657 (Other: World Health Organization (WHO))
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- People with Obesity: General population, respondents are recruited via email and/or phone through an online panel company with which respondents have provided permission to be contacted for research
  Interventions: Other: No treatment given
- Healthcare Providers: Health care professionals, respondents will be recruited via email, USPS mail, and/or phone through an online panel company with which respondents have provided permission to be contacted for research purposes or through the AMA Masterfile
  Interventions: Other: No treatment given
- Employer representatives: Employers, respondents will be recruited via email, USPS mail, and/or phone through an online panel company with which respondents have provided permission to be contacted for research purposes
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Completion of a questionnaire

SUMMARY:
The ACTION (Awareness, Care, and Treatment In Obesity management) study aims to identify perceptions, attitudes, behaviours, and potential barriers to effective obesity care across three respondent types: 1) People with Obesity, 2) Healthcare Providers and 3) Employer Representatives in the US. Data is collected via online surveys using a cross-sectional, US-based stratified sample design.

ELIGIBILITY:
Inclusion Criteria:

* GENERAL POPULATION
* Agrees to AE reporting
* Age at least 18 years
* Lives in the US
* Current BMI at least 30 kg/sqm
* HEALTH CARE PROFESSIONALS
* Agrees to AE reporting
* Physician and board certified or NP/PA
* Facility located in the U.S. and not Vermont
* Spends at least 70% of time in direct patient care
* Seen at least 100 patients in past month
* Seen at least 10 patients in past month needing weight management
* In practice 2-35 years
* Not competitively employed
* Primary Care Providers
* Specialty is FP, IM, GP
* Less than 50% patients seen for obesity
* Obesity Specialists
* Obesity medicine or weight loss specialist or at least 50% of patients seen for obesity
* In practice 2-35 years
* EMPLOYERS
* Age at least 18 years
* Works in the US
* Director, Administrator, CHRO, VP or other title
* Responsible for making or influencing decisions about health insurance or health and wellness programs
* Company employs 500 or more full-time employees
* Believes there is a weight issue at their company
* Not competitively employed

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 3767 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2015-11-12 (Actual); Study Completion 2015-11-12 (Actual)

PRIMARY OUTCOMES:
Awareness with the care and management of obesity among people with obesity | Start of interviews day 1 until day 15
  Data is collected via online questionnaires using a cross-sectional, US-based stratified sample design
Awareness with the care and management of obesity among health care providers | Start of interviews day 1 until day 15
  Data is collected via online questionnaires using a cross-sectional, US-based stratified sample design
Awareness with the care and management of obesity among employer representatives | Start of interviews day 1 until day 15
  Data is collected via online questionnaires using a cross-sectional, US-based stratified sample design

CONTACTS AND LOCATIONS:
Locations (1):
- Novo Nordisk Investigational Site, Honeoye Falls, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Result] Kaplan LM, Golden A, Jinnett K, Kolotkin RL, Kyle TK, Look M, Nadglowski J, O'Neil PM, Parry T, Tomaszewski KJ, Stevenin B, Lilleore SK, Dhurandhar NV. Perceptions of Barriers to Effective Obesity Care: Results from the National ACTION Study. Obesity (Silver Spring). 2018 Jan;26(1):61-69. doi: 10.1002/oby.22054. Epub 2017 Oct 31. PMID 29086529
- [Result] Jinnett K, Kyle T, Parry T, Stevenin B, Ramasamy A; ACTION Steering Group. Insights into the Role of Employers Supporting Obesity Management in People with Obesity: Results of the National ACTION Study. Popul Health Manag. 2019 Aug;22(4):308-314. doi: 10.1089/pop.2018.0133. Epub 2018 Oct 31. PMID 30383482
- [Result] Look M, Kolotkin RL, Dhurandhar NV, Nadglowski J, Stevenin B, Golden A. Implications of differing attitudes and experiences between providers and persons with obesity: results of the national ACTION study. Postgrad Med. 2019 Jun;131(5):357-365. doi: 10.1080/00325481.2019.1620616. Epub 2019 Jun 3. PMID 31155994
- [Derived] Dhurandhar NV, Kyle T, Stevenin B, Tomaszewski K; ACTION Steering Group. Predictors of weight loss outcomes in obesity care: results of the national ACTION study. BMC Public Health. 2019 Oct 30;19(1):1422. doi: 10.1186/s12889-019-7669-1. PMID 31666040